CLINICAL TRIAL: NCT04634396
Title: Telephone Acceptance and Commitment Therapy Intervention for Caregivers of Adults With Alzheimer's Disease and Related Dementias. A Single Arm Pilot
Brief Title: Possible Therapy by Phone for Caregivers
Acronym: TACTICs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Regenstrief Institute, Inc. (Other)
Responsible Party: Principal Investigator, Nicole R. Fowler, PhD, Associate Professor of Medicine, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 1904631305
Record Dates: First submitted 2020-11-03; First posted 2020-11-18 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Anxiety; Anxiety Disorders and Symptoms; Caregiver Burnout
Keywords: Alzheimer's disease; Dementia; Caregiving; Caregiver; Anxiety; Acceptance and commitment therapy; Telehealth
MeSH Terms: conditions — Anxiety Disorders; Caregiver Burden; Alzheimer Disease; Dementia

STUDY DESIGN:
Intervention Model Description: single arm proof of concept study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental TACTICs (Other): Telephone Acceptance and Commitment Therapy Intervention for Caregivers of adults with dementia (TACICS. Participants will receive a manualized acceptance and commitment therapy intervention delivered via phone in 6 weekly 1 hour sessions by a trained interventionalist
  Interventions: Behavioral: ACT Acceptance and Commitment Therapy

INTERVENTIONS:
Behavioral: ACT Acceptance and Commitment Therapy — 6 weeks of 1 hour sessions with a masters prepared research specialist to deliver validated tools

SUMMARY:
Caregivers of adults with dementia report higher stress, including anxiety and depressive symptoms, burden, and existential suffering, than caregivers of people with other chronic diseases.

DETAILED DESCRIPTION:
Acceptance and Commitment Therapy (ACT) is a behavioral intervention designed to increase psychological flexibility in the face of challenges. The Investigators are trying to determine proof of concept that suggests that ACT is effective in reducing anxiety and associated psychological distress in dementia caregivers. This study will recruit N=20 dementia caregivers to receive 6 weekly 1-hour telephone-based ACT sessions

ELIGIBILITY:
Inclusion Criteria:

* 21 years or older
* Able to communicate in English
* Able to provide informed consent
* Listed as primary caregiver in the chart of a patient with Alzheimer's disease or related dementia (DARD)
* Intends to continue caregiving form ADRD patient for at least 12 months or greater
* Clinically elevated anxiety score (score of 10 or higher on GAD-7)

Exclusion Criteria:

* Non-family member of the ADRD patient
* Has ADRD or other serious mental illness diagnosis such as bipolar or schizophrenia as determined by ICD-10 code

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-06-14 (Actual); Primary Completion 2019-12-09 (Actual); Study Completion 2019-12-09 (Actual)

PRIMARY OUTCOMES:
Anxiety symptoms measured by the Generalized Anxiety Disorder Scale (GAD-7) | through study completion, an average of 6 months
  Anxiety will be measured using the GAD-7 which contains 7 items with total scores ranging from 0 to 21. Scores of 5, 10 and 15 are cut off scores for mild, moderate and severe anxiety respectively. An add-on item assessing the patient's global impression of symptom related impairment helps researchers understand the extent to which anxiety interferes in daily life. The GAD-7 has factorial validity for the diagnosis of general anxiety disorder and is sensitive to change

SECONDARY OUTCOMES:
Depressive symptoms measured by the Patient Health Questionnarie-9 (PHQ-9) | through study completion, an average of 6 months
  Depressive symptoms will be measured using the 9 item Patient Health Questionnaire-9 (PHQ-9) to assess depressive symptoms. With total scores ranging from 0-27. scores of 5, 10, 15 and 20 represent mild, moderate, moderately severe and severe depression, respectively. The PHQ-9 has factorial validity for the diagnosis of major depressive disorder
Caregiver burden measured by the Zarit Burden Interview (ZBI) | through study completion, an average of 6 months
  Caregiver burden will be measured using the ZARIT Burden Interview (ZBI). This two
  factor 22 item scale measures personal strain and role strain in caregiving by summing
  responses to a total score (0-20) little or no burden; 21-40 mild to moderate burden; 41-60
  moderate to severe burden; and 61-88; severe burden). The ZBI measures change over time resulting from the progression of the patient's symptoms or from interventions aimed at reducing burden
Physical, emotional and existential suffering to caregivers measured by the Experience of Suffering Scale (ESS) | through study completion, an average of 6 months
  Well being will be measured using the (ESS). With prior testing in ADRD caregivers, the ESS contains 33 items across 3 subscales: physical (9items), psychological (15 items), and existential (9 items) suffering. Total scores for each subscale are calculated with higher scores indicating more suffering within each domain
Different strategies that caregivers use to cope measured with the Brief COPE | through study completion, an average of 6 months
  Coping will be measured with the 28 item Brief COPE. A measure of coping strategies used in response to stressors. Comprised of 28 coping strategies, the Brief COPE contains 14 two item subscales, each analyzed separately; self distraction, active coping, denial, substance use, use of emotional support, use of instrumental support, venting, behavioral disengagement, positive reframing, planning, humor, acceptance, religion and self-blame
Caregivers psychological flexibility measured by the Acceptance and Action Questionnaire-II (AAQ-II) | through study completion, an average of 6 months
  Psychological flexibility and its opposite, experiential avoidance will be measured using the 7 item Acceptance and Action Questionnaire-II (AAQ-II). Respondents rate how true each statement (e,g it is okay if I remember something unpleasant) is for them on a 7 point Likert type scale anchored from 1=never true to 7- always true. Higher scores indicate greater psychological flexibility or acceptance
Overall quality of life will be measured with the NIH PROMIS Global Health measure | through study completion, an average of 6 months
  Quality of Life will be assessed with the 10-item PROMIS Global Health measure. On a 5-point scale, participants rate their mental and physical well-being with higher scores indicative of better health
Caregivers grief during active caregiving will be measured with the Anticipatory Grief Scale (AGS) | through study completion, an average of 6 months
  Anticipatory grief will be measured by the AGS, a 27 item self report tool designed to assess the bereavement experience of dementia caregivers. Items are scored on a 5-point Likert type scale with responses ranging from "strongly disagree" to "strongly agree".

OTHER OUTCOMES:
The feasibility of the TACTICs Intervention will be measured by accrual rate, attendance of sessions, and the retention in the study | baseline and through study completion, an average of 6 months.
  The investigators will assess the number of eligibly screened caregivers who choose to consent and enroll in the pilot study, assess the total number of sessions that participants attend the number of enrolled subjects completing the outcome assessments.
Caregivers acceptability of the TACTICs intervention | through study completion, an average of 6 months
  The investigators will assess intervention acceptability using a brief investigator created battery of qualitative and quantitative satisfaction items

CONTACTS AND LOCATIONS:
Overall Officials: Shelley A. Johns, PhD, Principal Investigator — Indiana University
Locations (1):
- Regenstrief Institute, Inc., Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
In future manuscripts, the authors will list contact information and state that IPD is available upon request
Time Frame: Spring, 2021
Access Criteria: manuscripts